CLINICAL TRIAL: NCT02879253
Title: Evaluation of Inter-patient Variability Size of the Nasal Cavity, Based on CT Scans
Acronym: NEMROfentes3D
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2015/280
Record Dates: First submitted 2016-08-10; First posted 2016-08-25 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Nasal Cavity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is part of the french research program ANR NEMRO "MICROROBOTIC NASAL ENDOSCOPY BY OPTICAL COHERENCE TOMOGRAPHY: IMPACT OF SMELL DEFICIENCY ON NEURODEGENERATIVE DISEASES." Recent studies have shown a strong correlation between the decrease in olfactory faculties of patients and the presence of neurodegenerative diseases.

This possible relationship has created a need to inspect in detail the area of the nasal cavity that houses the olfactory function.

Thus, the purpose of NEMRO project is developing a robot to explore olfactory slots of patients, with a view to extract images through non invasive imaging probe, and hoping to identify early signs of degeneration the olfactory tissue. The robot developed will thus be able to navigate in the nasal cavity of patients, and to break into the olfactory slots, which will host the imaging phase.

The purpose of this study is therefore to collect data on the usual path of instruments (endoscope, for example) in this area, and future potential pathway of the robot. This collection made from Computed Tomography (CT) scans will define the clinical geometry of the target area and provide precisely the dimensional constraints needed to build the NEMRO robot .

ELIGIBILITY:
Inclusion Criteria:

* men or women aged >18

Exclusion Criteria:

* any pathology observed on the scan (sinusitis, cancer, previous surgery ...), that could interfere with the evaluated parameters, according to the medical expert

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CT scans of men and women > 18 years will be observed. Age selected corresponds to a period where the nasal cavity is completely formed, with no more structural and morphological changes due to the growth of the individual in the development phase; regarding sex study subjects, an equal distribution between men and women is required wherever possible.
  Will be excluded images suggesting a pathology that could interfere with the target parameters of the study in the area, according to the opinion of the maxillofacial surgeon in charge of the collection (sinusitis, cancer, previous surgery ...).
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-12-24 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2016-07-11 (Actual)

PRIMARY OUTCOMES:
Width of the nasal cavity and olfactory slots | at enrollment
  Distance measurements to evaluate the width of the nasal cavity and olfactory slots, on previous available imaging. Composite primary outcome.
Geometry of the nasal cavity and olfactory slots | at enrollment
  Assesment of the geometry of the nasal cavity and olfactory slots, on previous available imaging. Composite primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No